CLINICAL TRIAL: NCT07043413
Title: Thrombus Analysis of Ischemic Stroke
Acronym: TAOIST
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Min Kim, Professor, Seoul National University Hospital
Other Study IDs: TAOIST
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction; thrombus; stroke mechanism; prognosis
MeSH Terms: conditions — Cerebral Infarction; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human thrombus obtained after endovascular thrombectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thrombus analysis — Detailed expression pattern of RNA and histological characteristics will be investigated.

SUMMARY:
Patients with acute ischemic stroke who have undergone endovascular thrombectomy will be eligible to be included, and thrombus will be collected after obtaining informed consent. Enrolled patients will receive a comprehensive diagnostic evaluation and the best medical treatment according to recent stroke management guidelines. The mechanism of the stroke will be classified into atherosclerotic, cardiac embolism, others and unknown causes based on diagnostic workup. Patients will be monitored in an outpatient clinic for vascular events including stroke recurrence, death, and bleeding events, which will continue for up to two years after the initial stroke event. Thrombus information related to RNA expression patterns and histological characteristics will be analyzed to classify the stroke mechanism and predict future vascular events after the initial stroke.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute ischemic stroke who had undergone endovascular thrombectomy

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with acute ischemic stroke who had undergone endovascular thrombectomy and agreed to participate to the study
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular events | two years after initial stroke
  major vascular events after endovascular thrombectomy, including stroke, myocardial infarction, and vascular death

SECONDARY OUTCOMES:
Thromboembolic events | two years after initial stroke
  Any thromboembolic events after endovascular thrombectomy including ischemic stroke, transient ischemic attack, myocardial infarction or unstable angina, peripheral artery disease requiring hospitalization, venous thromboembolism, pulmonary embolism and vascular death

OTHER OUTCOMES:
overall mortality | two years after initial stroke
  any death event after endovascular thrombectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jong-ro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided